CLINICAL TRIAL: NCT00126568
Title: Phase II Trial of BAY 43-9006 in Patients With Advanced Anaplastic Carcinoma of the Thyroid
Brief Title: Sorafenib in Treating Patients With Advanced Anaplastic Thyroid Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00118; NCI-2009-00118 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 5304; CDR0000437789; CASE 5304 (Other: Case Western Reserve University); 7037 (Other: CTEP); U01CA062502 (NIH)
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Results first posted 2012-08-10 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: Anaplastic Thyroid Cancer; Recurrent Thyroid Cancer
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic; Thyroid Neoplasms | interventions — Sorafenib

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN

SUMMARY:
This phase II trial is studying how well sorafenib works in treating patients with advanced anaplastic thyroid cancer. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine whether the objective response rate is ≥ 20% in patients with advanced anaplastic thyroid cancer treated with sorafenib.

II. Determine the survival of patients treated with this drug. III. Determine the safety profile of this drug in these patients. IV. Determine the pharmacokinetic predictors of response to this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed for survival.

ELIGIBILITY:
Criteria:

* Progressive disease after prior cytotoxic chemotherapy (i.e., chemotherapy alone or combined with radiotherapy)
* No symptomatic bulky disease that would impair the airway or impede swallowing (for patients with ECOG performance status 2)
* No known brain metastases
* Measurable or evaluable disease

  * Measurable disease, defined as ≥ 1 unidimensionally measurable lesion >= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan
  * Measurable disease not in a previously irradiated field
* Patients with evidence of abnormal cardiac conduction (e.g., bundle branch block or heart block) are eligible provided disease has been stable for the past 6 months
* Performance status:

  * ECOG 0-2 OR Karnofsky 50-100%
* Life expectancy more than 8 weeks
* Absolute neutrophil count >= 1,250/mm3
* Platelet count >= 100,000/mm3
* No evidence of bleeding diathesis
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* PTT =< 1.5 times ULN
* Creatinine =< 1.5 times ULN
* No myocardial infarction within the past 6 months
* No New York Heart Association class III or IV cardiac disease
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No uncontrolled hypertension (i.e., systolic blood pressure (BP) > 150 mm Hg OR diastolic BP > 100 mm Hg)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow oral medication
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to sorafenib
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No other uncontrolled illness
* No more than 2 prior systemic cytotoxic chemotherapy regimens (combined modality systemic cytoxic chemotherapy is considered 1 prior cytotoxic regimen)
* At least 7 days since prior chemotherapy and recovered
* At least 7 days since prior radiotherapy and recovered
* No prior sorafenib or other inhibitors of MAP kinase signaling intermediates
* No prior cancer treatment that would preclude study participation
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No concurrent cytochrome P450 enzyme-inducing antiepileptic drugs (e.g., phenytoin, carbamazepine, or phenobarbital)
* No concurrent Hypericum perforatum (St. John's wort) or rifampin
* No concurrent therapeutic anticoagulation (concurrent prophylactic anticoagulation (i.e., low-dose warfarin) for venous or arterial access devices allowed provided requirements for INR and PTT are met)
* No other concurrent anticancer therapy
* Histologically confirmed anaplastic* thyroid cancer

  * Not amenable to definitive curative surgery or radiotherapy [Note: *Papillary, follicular, or other histologies that are mixed or identified in a diagnostic tissue sample are allowed provided a high-grade undifferentiated anaplastic component is present ]
* No cardiac arrhythmia
* AST and ALT =< 3.5 times ULN
* INR < 2.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panayiotis Savvides, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Savvides P, Nagaiah G, Lavertu P, Fu P, Wright JJ, Chapman R, Wasman J, Dowlati A, Remick SC. Phase II trial of sorafenib in patients with advanced anaplastic carcinoma of the thyroid. Thyroid. 2013 May;23(5):600-4. doi: 10.1089/thy.2012.0103. Epub 2013 Apr 18. PMID 23113752

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from June 2005 to April 2011 from medical clinics
Groups:
- BAY 43-9006: BAY 43-9006 (sorafenib) will be administered on a fixed daily oral dosing schedule of 400 mg twice daily. A cycle of therapy will be considered 28 days (4 weeks / 1 month).
Period: Overall Study
Arm/Group | BAY 43-9006
Started | 20
Completed | 18 (Disease progression at beginning of study, not evaluable)
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | BAY 43-9006
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 59 [28 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Response to Treatment Measured by RECIST Criteria
Description: Response evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. The patient's best response depends on the achievement of measurement and confirmation criteria of Complete Response (CR), Stable Disease (SD), Partial Response (PR) or Progressive Disease (PD). Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques (CT, MRI, x-ray) or as >10 mm with spiral CT scan.
Time Frame: at 6 months after treatment
Population: All patients that received at least one cycle of treatment
Measure: Number; unit: participants
Arm/Group | BAY 43-9006
Number analyzed (Participants) | 18
participants
  Partial Response | 2
  Stable Disease | 5
  Progressive Disease | 11

2. Secondary Outcome: Progression Free Survival Was Measured From the Date of Outset of Treatment to the Date of Disease Progression.
Time Frame: 27 months
Population: All patients on study
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BAY 43-9006
Number analyzed (Participants) | 20
months | 1.9 [1.3 to 3.6]

3. Secondary Outcome: Overall Survival Was Measured From the Date of Outset of Treatment to the Date of Death.
Time Frame: 27 months
Population: All patients on study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BAY 43-9006
Number analyzed (Participants) | 20
months | 3.9 [2.2 to 7.1]

4. Secondary Outcome: Number of Participants That Experienced Adverse Events to Characterize the Safety Profile of BAY 43-9006
Description: The safety and toxicity profile of BAY 43-9006 as measured by toxicity grades of adverse events.
Time Frame: 27 months
Population: Any participant that received treatment was analyzed for adverse events. Detailed information is reported in the Adverse Events data table.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sorafenib Tosylate)
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Time Frame: Adverse events were collected weekly for the duration that the patients started on treatment to end of study.
Arm/Group | BAY 43-9006
Serious Adverse Events (participants affected / at risk) | 8/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAY 43-9006 (N=20)
Death not associated with CTCAE term - Death NOS(not otherwise specified) (General disorders) | 1 (1)
Death not associated with CTCAE term - Disease progression NOS(not otherwise specified) (General disorders) | 3 (3)
Death not associated with CTCAE term - Sudden death (General disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (7)
Edema: limb (Blood and lymphatic system disorders) | 1 (2)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1 (1)
Infection with unknown ANC(Absolute neutrophil count) - Lung (pneumonia) (Infections and infestations) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2)
Pain - Abdomen NOS(not otherwise specified) (Gastrointestinal disorders) | 1 (1) — NOS- not otherwise specified
Pain - Eye (Eye disorders) | 1 (2)
Perforation, GI - Appendix (Gastrointestinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAY 43-9006 (N=20)
ALT(Alanine transaminase), SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 3 (8)
AST(aspartate aminotransferase), SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 4 (7)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 8 (22)
Alkaline phosphatase (Metabolism and nutrition disorders) | 4 (4)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 6 (6)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 2 (2)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 2 (2)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (3)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 8 (34)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Cardiac troponin I (cTnI) (Cardiac disorders) | 1 (1)
Cervical spine-range of motion (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (8)
Constitutional Symptoms - Other (Specify, __) (General disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Creatinine (Metabolism and nutrition disorders) | 4 (6)
Dehydration (Gastrointestinal disorders) | 1 (1)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 9 (20)
Distension/bloating, abdominal (Gastrointestinal disorders) | 2 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (7)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 7 (9)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Edema: head and neck (Blood and lymphatic system disorders) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 14 (18)
Fever (in the absence of neutropenia) (General disorders) | 2 (2) — Where neutropenia is defined as Absolute Neutrophil Count (ANC) <1.0 x 10e9/L)
Flushing (Skin and subcutaneous tissue disorders) | 5 (6)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 10 (28)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 2 (4)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 5 (5)
Hemoglobin (Blood and lymphatic system disorders) | 14 (33)
Hemorrhage, GI - Lower GI NOS(not otherwise specified) (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GI - Oral cavity (Gastrointestinal disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory - Bronchopulmonary NOS(not otherwise specified) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory - Larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory - Respiratory tract NOS(not otherwise specified) (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Cardiac disorders) | 4 (5)
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 2 (5)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1 (1)
Infection with normal ANC(Absolute Neutrophil Count) or Grade 1 or 2 neutrophils - Pharynx (Infections and infestations) | 1 (1)
Infection with normal ANC(Absolute Neutrophil) or Grade 1 or 2 neutrophils - Upper aerodigestive NOS (Infections and infestations) | 1 (1)
Infection with normal ANC(Absolute Neutrophil Count) or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 2 (2)
Infection with normal ANC(Absolute Neutrophil Count) or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 1 (1)
Infection with normal ANC(Absolute Neutrophil Count) or Grade 1 or 2 neutrophils - Vagina (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Leukocytes (total White Blood Count) (Blood and lymphatic system disorders) | 7 (9)
Lymphopenia (Blood and lymphatic system disorders) | 16 (77)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 (2)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 (4)
Mood alteration - Depression (Nervous system disorders) | 1 (1)
Mucositis/stomatitis (clinical exam) - Oral cavity (General disorders) | 7 (7)
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 4 (11)
Neurology - Other (Specify, __) (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 8 (9)
Neutrophils/granulocytes (ANC(absolute neutrophil count)/AGC(absolute granulocyte count) (Blood and lymphatic system disorders) | 2 (8)
Obstruction/stenosis of airway - Trachea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 1 (1)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 3 (5)
Pain (General disorders) | 3 (3)
Pain - Abdomen NOS (not otherwise specified) (General disorders) | 1 (4)
Pain - Back (General disorders) | 6 (7)
Pain - Chest/thorax NOS (not otherwise specified) (General disorders) | 8 (9)
Pain - Extremity-limb (General disorders) | 2 (4)
Pain - Face (General disorders) | 1 (1)
Pain - Head/headache (General disorders) | 4 (5)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 2 (4)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain - Neck (General disorders) | 2 (2)
Pain - Oral cavity (General disorders) | 2 (2)
Pain - Pelvis (General disorders) | 2 (2)
Pain - Scrotum (General disorders) | 1 (1)
Pain - Stomach (General disorders) | 1 (1)
Pain - Throat/pharynx/larynx (General disorders) | 4 (4)
Pain - Tumor pain (General disorders) | 1 (1)
Pain-Eye (Eye disorders) | 1 (1)
Perforation, GI - Appendix (Gastrointestinal disorders) | 1 (1)
Pericardial effusion (non-malignant) (Cardiac disorders) | 2 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 5 (9)
Platelets (Blood and lymphatic system disorders) | 4 (5)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 (23)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3 (3)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 10 (23)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash: dermatitis associated with radiation - Chemoradiation (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: dermatitis associated with radiation - Radiation (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 6 (13)
Rigors/chills (General disorders) | 2 (3)
Salivary gland changes/saliva (Gastrointestinal disorders) | 1 (1)
Secondary Malignancy - possibly related to cancer treatment (Specify, __) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 11 (22)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 (2)
Stricture/stenosis (including anastomotic), GI - Pharynx (Gastrointestinal disorders) | 1 (1)
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 6 (9)
Sweating (diaphoresis) (General disorders) | 2 (2)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 1 (1)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 5 (5)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1)
Vision-flashing lights/floaters (Eye disorders) | 1 (1)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Vomiting (Gastrointestinal disorders) | 2 (10)
Weight loss (Investigations) | 9 (15)

LIMITATIONS AND CAVEATS:
The study met the pre-specified criteria for enrollment of all planned 32 patients. However due to poor accrual the study was halted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less